CLINICAL TRIAL: NCT02715934
Title: Glucose to Goal: A Model to Support Diabetes Management in Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Linda Siminerio, Professor of Medicine, University of Pittsburgh
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1R34DK106684-01A1 (NIH)
Record Dates: First submitted 2016-03-01; First posted 2016-03-22 (Estimated); Last update posted 2018-04-10 (Actual); Status verified 2018-04

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes Education; Chronic Disease Management; Health Care Delivery; Patient-Centered Medical Home; Primary Care
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Glucose to Goal (Experimental): Three diabetes educators will be assigned to the Glucose to Goal/experimental arm. The educators will each identify two primary care practices of mid to large size to participate in the Glucose to Goal intervention. Patients will not be formally recruited or enrolled. Rather, information documented in the electronic medical record system will be extracted to evaluate patient-level outcomes. Based on a random sampling of mid to large size primary care practices in study communities, an estimated 2,200 patients with diabetes per study group will meet eligibility criteria for DSME referral.
  Interventions: Other: Glucose to Goal
- Control Group (Other): Two usual care diabetes educators will each identify three primary care practices of mid to large size to include in the control arm and participate in the usual care intervention. Uneven group assignment accounts for the amount of time (one day equivalent/per week) that the intervention diabetes educators will devote to each primary care practice versus the full-time availability of the usual care diabetes educators to see patients at the outpatient, hospital-based program. Like the experimental arm, an estimated 2,200 patients with diabetes will meet eligibility criteria for DSME referral. Patients will not be formally recruited or enrolled into the control arm; data will be extracted from the electronic medical record system to evaluate patient-level outcomes.
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Glucose to Goal — The Glucose to Goal intervention applies elements of the Patient Centered Medical Home (i.e., practice design, decision support, population management, etc) to diabetes education services and operationalizes the current DSME objectives in the primary care setting.
  Arms: Glucose to Goal
Other: Usual Care — The control group will follow the traditional DMSE delivery model, which includes primary care providers referring patients to an outpatient, hospital-based diabetes educator for DSME, but in a passive manner (i.e., without proactive patient identification), which is the usual process for referrals.
  Arms: Control Group

SUMMARY:
Diabetes education is a very important part of diabetes care. Most people with diabetes receive care in primary care practices where diabetes education is not always available. This project tests a model designed to improve access to diabetes education services.

DETAILED DESCRIPTION:
Evidence that diabetes self-management education (DSME) can improve health outcomes has repeatedly been shown and is considered to be a critical component of care. Diabetes educators are highly skilled at addressing diabetes-related clinical and behavioral needs through DSME, but engagement with diabetes educators is underutilized. It has been suggested that poor referral practices and the way in which DSME service is delivered are the problems. Most patients receive diabetes care in primary care yet most DSME programs are distinctly separate from primary care practice. This limits care coordination and diabetes educator access to amenities currently available to primary care. Efforts are underway to change the US health care paradigm with a focus on quality in primary care that includes practice redesign, population management, and communication through electronic medical records. The purpose of this application is to evaluate the deployment of Glucose to Goal, a model relying on a systematic redesign of practice that links diabetes educators services with primary care. This will be compared to the traditional process for DSME delivery, without the direct connection to primary care processes, for an eighteen month period. The hypothesis is that the proportion of primary care provider referrals and patient utilization of diabetes educator services from primary care practices participating in Glucose to Goal will be higher compared to those associated with traditional DSME. It is anticipated that this model will appeal to primary care providers, demonstrate a feasible approach to offering diabetes education in the current health environment, and set the stage for future testing of the model, namely its impact on meaningful improvements on diabetes outcomes and cost-effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of type 2 diabetes
* Patients referred to diabetes self-management education by their primary care provider
* Able to read and write English

Exclusion Criteria:

* Clinical diagnosis of type 1 or gestational diabetes
* Unable to speak or read English

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4994 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Provider referral | Monitor continuously across 18 months
  The proportion of provider referrals for DSME divided by the total number of patients eligible for a referral. Patients will be considered eligible for referral if they were seen by their primary care provider during the intervention period and the provider did not contraindicate DSME for any reason. Referrals (eligibility for and made) will be tracked through electronic medical record review.

SECONDARY OUTCOMES:
Patient participation | Monitor continuously across 18 months
  Patient participation will be reported as the proportion of patients who participate in DSME divided by the total number of eligible patients from each participating primary care practice during the study period and will take into account patterns and frequency of visits. Patients will be considered eligible if they have received a referral to DSME from their primary care provider. Patients will be offered the opportunity to meet with the diabetes educator for a series of DSME visits and these visits will occur in individual or group format, depending on space, scheduling, etc. The number and content of the visits will be patient-centered (driven by the patient). Patients eligible for and participating in DSME will be tracked through electronic medical record review.

OTHER OUTCOMES:
Primary care practice satisfaction with implementation process | Baseline, 9 months, 18 months
  The research team will collect data on the implementation process at the primary care practice orientation and team huddles at the mid-point and end of the intervention. During the practice orientation, the manner in which practices negotiate adoption of the key features of Glucose to Goal will be documented. With the assistance of trained qualitative researchers, mid and end point team huddles will be conducted using a focus group format to review experiences, examine challenges and barriers, identify best practices, and gauge provider and diabetes educator satisfaction.
Hemoglobin A1c | As available across 18 months
  In preparation for a larger scale, longitudinal study testing the effectiveness of the Glucose to Goal model on diabetes control, hemoglobin A1c values and other key diabetes markers (i.e., lipid panels, blood pressure) that are documented in the electronic medical record system during the study period will be extracted and analyzed. Dates and frequency of tests, absolute values, and whether values were within recommended target ranges will be documented.
Problem Assessment in Diabetes-5 (PAID-5) | As available across 18 months
  PAID is a measure of psychosocial adjustment and diabetes emotional distress. Psychometric reports to date on PAID have shown it to have consistently high internal and test-retest reliability; correlate strongly with a wide range of theoretically related constructs such as general emotional distress, depression, diabetes self-care behaviors, diabetes coping, and health beliefs; and be a statistically significant predictor of glycemic control (Polonsky et al, 1995). The 5-item version (McGuire et al, 2010) will be administered at DSME visits.
Diabetes Empowerment Scale - Short Form (DES-SF) | As available across 18 months
  To allow for a brief overall assessment of diabetes-related psychosocial self-efficacy, the DES-SF, an 8-item scale, was developed based on the original 37-item DES (Anderson et al, 2003). DES-SF items address participants' perceived ability to assess readiness to change, set/reach goals, overcome barriers, cope with emotions, manage stress, obtain support, motivation, and make cost/benefit decisions. The DES-SF will be administered at DSME visits.
Summary of Diabetes Self-care Activities Measure (SDSCA) | As available across 18 months
  This instrument will be used to evaluate self-care with questions about number of days in a week that the participant reports self-care behaviors related to general diet, specific diet, exercise, blood glucose testing, foot care, and smoking. Correlations with other measures of diet and exercise generally support validity of SDSCA subscales (Toobert et al, 2000). The SDSCA will be administered at DSME visits.

CONTACTS AND LOCATIONS:
Overall Officials: Linda Siminerio, RN, PhD, CDE, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Community Medicine, Inc., Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] Polonsky WH, Anderson BJ, Lohrer PA, Welch G, Jacobson AM, Aponte JE, Schwartz CE. Assessment of diabetes-related distress. Diabetes Care. 1995 Jun;18(6):754-60. doi: 10.2337/diacare.18.6.754. PMID 7555499
- [Background] McGuire BE, Morrison TG, Hermanns N, Skovlund S, Eldrup E, Gagliardino J, Kokoszka A, Matthews D, Pibernik-Okanovic M, Rodriguez-Saldana J, de Wit M, Snoek FJ. Short-form measures of diabetes-related emotional distress: the Problem Areas in Diabetes Scale (PAID)-5 and PAID-1. Diabetologia. 2010 Jan;53(1):66-9. doi: 10.1007/s00125-009-1559-5. Epub 2009 Oct 20. PMID 19841892
- [Background] Anderson RM, Fitzgerald JT, Gruppen LD, Funnell MM, Oh MS. The Diabetes Empowerment Scale-Short Form (DES-SF). Diabetes Care. 2003 May;26(5):1641-2. doi: 10.2337/diacare.26.5.1641-a. No abstract available. PMID 12716841
- [Background] Toobert DJ, Hampson SE, Glasgow RE. The summary of diabetes self-care activities measure: results from 7 studies and a revised scale. Diabetes Care. 2000 Jul;23(7):943-50. doi: 10.2337/diacare.23.7.943. PMID 10895844
- [Derived] Krall JS, Kanter JE, Ruppert KM, Arena VC, Solano FX, Siminerio LM. Effect of a Primary Care-Based Diabetes Education Model on Provider Referrals and Patient Participation. Sci Diabetes Self Manag Care. 2021 Feb;47(1):74-84. doi: 10.1177/0145721720981840. PMID 34078203